CLINICAL TRIAL: NCT02570776
Title: Prevalence of Helicobacter Pylori Infection in Dyspeptic Adults and Validation of C14 Urea Breath Test (UBT) as a Diagnostic Tool for Helicobacter Pylori Infection in Pakistani Population
Brief Title: UBT as a Diagnostic Tool for HP Prevalance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Liver & GI Diseases, Pakistan (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Dr. Zahid Azam, Professor Medicine & Gastroenterology, National Institute of Liver & GI Diseases, Pakistan
Other Study IDs: PK-13-01
Record Dates: First submitted 2014-05-07; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Dyspepsia
Keywords: Helicobacter pylori; UBT; Sensitivity; specificity; prevalence
MeSH Terms: conditions — Dyspepsia; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation: Cohort of patients for Endoscopy & they are assessed for Helicobacter pylori through the histopathology & also throgh C14 C UBT.

SUMMARY:
The prevalence of H. pylori infection in Pakistan is unknown and investigators want to assess it in dyspeptic patients utilizing UBT. At the same time investigators want to validate UBT sensitivity and specificity in Pakistani patients

DETAILED DESCRIPTION:
The non-invasive methods for the diagnosis of Hp are the Urea Breath Test (UBT) and serological tests. The serological tests includes ELISA test in serum for Hp antibody and in stool for Hp antigen. Serum ELISA Hp antibody is not sensitive for showing active infection and the titres do not decrease even after successful eradication. Serology test cannot be used for those who have previously been treated for Hp, as the decline in titre of Hp antibodies is too slow to be of practical use. The stool Hp antigen detection test is more sensitive and specific as it detects bacterial antigens which will only be positive in the presence of Hp. However, it is cumbersome to collect stool and laboratory services are required. The C14 Urea Breath Test (UBT) is an office based test with sensitivity and specificity comparable to that of the stool antigen test. The diagnostic validity of these tests depends on the prevalence of H pylori infection. A higher prevalence would be associated with higher sensitivity and lower specificity. The safety profile of the urea breath test is very favourable, and no major side effects are associated with it. The aims of this study are to estimate H pylori prevalence in Pakistan among the adult dyspeptic population and to validate the sensitivity and specificity UBT in our population

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with dyspeptic symptoms (B1 Criteria of FD)
* Subject who has not been treated for H pylori eradication in the past
* Age above 18 years
* No Alarm symptoms of :

  * Gastrointestinal Bleeding
  * Anemia
  * Early satiety
  * Unexplained weight loss
  * Progressive dysphagia
  * Odynophagia
  * Recurrent vomiting
  * Family history of GI malignancy
  * Previous GI malignancy

Exclusion Criteria:

* Pregnant females
* Use of NSAIDs
* Use of anti- secretory agent (H2 blockers) and proton pump inhibitors in previous 4 weeks
* Use of anti- microbial agents (Clarithromycin, Metronidazole, Amoxacillin, quinalones) or bismuth in last 4 weeks
* .Gastric and/or duodenal erosions or ulcers, polyps or malignancy if noted on endoscopy will be excluded.
* Patients with predominant symptoms or gastro esophageal reflux disease (GERD) or Endoscopic evidence of esophagitis.
* Patients with abnormal upper abdominal ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients getting routine upper GI Endoscopy are enrolled and as per routine histopathology samples are taken to assess Helicobacter pylori. This assessment will be done by two independent histopathologists & later the results will be compared with C14 UBT taking histopathology as gold standard.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of H pylori infection in Pakistani polulation | 1 day
  Prevalence of H pylori will be assessed by UBT & confirmed with histopathology as gold standard & sensitivity & specificity will be calculated.

SECONDARY OUTCOMES:
Sensivity & specificity of Heliprobe (C14 UBT system) in local population | 1 day
  Sensitivity & specificity will be measured by number of subjects positive based on ROC

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Azam, FCPS, MSc, Principal Investigator — National Institute of Liver & GI Diseases, Dow University of Health Sciences
Locations (1):
- National Institute of Liver & GI Diseases, Dow University of Health Sciences, Karachi, Sindh, Pakistan